CLINICAL TRIAL: NCT05942391
Title: Fast Recovery from Anxiety-related Disorders: Brief-intensive CBT Versus Once-weekly CBT
Brief Title: Brief-intensive CBT Versus Once-weekly CBT in Anxiety-related Disorders
Acronym: KOMMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Free University Medical Center (Other)
Collaborators: Netherlands Brain Foundation (Other)
Responsible Party: Principal Investigator, Dr. Adrie Seldenrijk, Principal investigator, Free University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DR2022-00396
Record Dates: First submitted 2023-06-16; First posted 2023-07-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Anxiety Disorders; Obsessive-Compulsive Disorder; Posttraumatic Stress Disorder; Hypochondriasis
Keywords: agoraphobia; social anxiety disorder; generalized anxiety disorder; panic disorder; trauma; health anxiety; obsessive compulsive disorder; CBT
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic; Hypochondriasis; Agoraphobia; Phobia, Social; Generalized Anxiety Disorder; Panic Disorder; Wounds and Injuries | interventions — Cognitive Behavioral Therapy; Implosive Therapy

STUDY DESIGN:
Intervention Model Description: a parallel-group randomised controlled intervention study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief-Intensive CBT (Experimental): 16 sessions in 2 weeks + 4 follow up sessions. The CBT consists of 16 sessions exposure therapy, spread over 4 half-days in 2 weeks, + 4 sessions within 3 months.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- weekly CBT (Active Comparator): 20 weekly CBT sessions within 5 to 6 months. The CBT consists of exposure therapy.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — The intervention is brief-intensive, guided exposure therapy and consists of 16 sessions exposure therapy, spread over 4 half-days in 2 weeks plus 4 follow-up sessions within 3 months.
  Other Names: exposure therapy

SUMMARY:
The goal of this clinical trial is to compare brief-intensive cognitive-behaviour therapy (CBT) with regular weekly CBT in people with anxiety-related disorders.

The main question to answer is: will brief-intensive CBT improve functioning (work, family, social) more and faster than does regular weekly CBT?

Participants will be asked to follow CBT treatment (20 sessions of 45 minutes in both conditions), and participate in 7 measurements with a total duration of 5 hours over 1 year.

Researchers will compare:

* Brief-intensive CBT: 16 sessions in 2 weeks + 4 follow-up sessions within 3 months
* Regular CBT with 20 weekly sessions in 6 months

DETAILED DESCRIPTION:
Rationale: Anxiety-related disorders (i.e., obsessive compulsive, health anxiety and trauma disorders) affect about 10% of the adults. Though clinically heterogeneous, transdiagnostic aspects are expected disasters, anxiety and avoidance. Profound impairments include work and family functioning. Many enter a vicious circle with comorbidity and further decline in quality of life. Hence, the impact on functioning is tremendous, with anxiety-related disorders rating highest on disability rankings in the age 15-64 years. Cognitive behavioral therapy (CBT) is the preferred and often only psychotherapy for these disorders. Because guidelines are based on weekly sessions, recovery takes half a year at least. Based on initial research findings, we expect faster recovery by providing CBT in a brief-intensive format (BI-CBT), with clear benefts for patients, families and society. Some institutions already provide BI-CBT. However, evidence to justify this or to further implement BI-CBT is insufficient.

Study design: a parallel-group randomised controlled multicenter intervention study.

Study population: Adults aged 18-65 yr old with an anxiety-related disorder (panic, agrophobia, social anxiety, generalised anxiety obsessions/compulsions, health anxiety and post-traumatic stress)

Intervention (if applicable): One group receives BI-CBT (16 sessions in 2 weeks + 4 follow up sessions) and the other group receives 20 weekly CBT sessions. Treatment in both conditions can be personalised by a focus on work or family functioning.

Main study parameters/endpoints: The main study parameter is the 'area under the curve' for 6-month health and disability. Also, 1 year efficacy (both on functioning and symptom-level), cost-effectiveness, and feasibility will be assessed. Potential predictors of treatment preference, efficacy and drop-out will be explored.

All patients are expected to follow CBT (20 sessions of 45min) and participate in 7 measurements over 1 year.

The general measurements are online questionnaires and interviews by telephone, asking about someones functioning, quality of life and symptoms of anxiety or depression, how one copes with these and what one expects of the therapy.

The acronym KOMMA is based on the Dutch translation of 'to put a quick end to anxiety': Korte Metten Met Angst.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older;

Reaching out for mental health care for one of the following disorders:

panic disorder, agoraphobia, generalised anxiety disorder, social anxiety disorder, posttraumatic stress disorder, obsessive-compulsive disorder, health anxiety disorder.

Exclusion Criteria:

* Is in need of emergency mental health care
* Has insufficient language skills in Dutch
* Has evident cognitive limitations
* Has had changes in the use of medication during the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the health and disability Curve at 6 months | baseline, 2 weeks, 4 weeks, 2 months, 3 months, 6 months
  The 'area under the curve' for health and disability is based on the 36-item self-report World Health Organisation Disability Assessment Schedule (WHODAS 2.0). The WHODAS 2.0 captures the level of functioning in six domains of life: Cognition, Mobility, Self-care, Getting along, Life activities, Participation. Possible total scores of the items across all domains range 0 - 100. Lower scores indicate less disability.

SECONDARY OUTCOMES:
Area Under the health and disability Curve at 12 months | baseline, 2 weeks, 4 weeks, 2 months, 3 months, 6 months, 12 months
  The 'area under the curve' for health and disability is based on the 36-item self-report World Health Organisation Disability Assessment Schedule (WHODAS 2.0). The WHODAS 2.0 captures the level of functioning in six domains of life: Cognition, Mobility, Self-care, Getting along, Life activities, Participation. Possible total scores of the items across all domains range 0 - 100. Lower scores indicate less disability.
Change from baseline in severity of anxiety symptoms at post-treatment | baseline and 3 or 6 months
  Severity of anxiety-related disorder, measured with the following disorder-specific severity questionnaires: the 24-item Liebowitz Social Anxiety Scale self-report version, the 7-item Panic Disorder Severity Scale self-report version, the 28-item Mobility Inventory, the 16-item Penn State Worry Questionnaire, the 10-item Yale-Brown Obsessive Compulsive Scale self-report version, the 20-item PTSD checklist for the DSM-5, or the 14-item Whitely Index. Higher scores indicate higher symptom severity. Z-scores will be calculated from individual scores for group-level analyses.
Change from baseline in severity of anxiety symptoms at 3 months | baseline and 3 months
  Severity of anxiety-related disorder, measured with the following disorder-specific severity questionnaires: the 24-item Liebowitz Social Anxiety Scale self-report version, the 7-item Panic Disorder Severity Scale self-report version, the 15-item Fear Questionnaire, the 16-item Penn State Worry Questionnaire, the 10-item Yale-Brown Obsessive Compulsive Scale self-report version, the 20-item PTSD checklist for the DSM-5, or the 14-item Whitely Index. Higher scores indicate higher symptom severity. Z-scores will be calculated from individual scores for group-level analyses.
Change from baseline in severity of anxiety symptoms at 12 months | baseline and 12 months
  Severity of anxiety-related disorder, measured with the following disorder-specific severity questionnaires: the 24-item Liebowitz Social Anxiety Scale self-report version, the 7-item Panic Disorder Severity Scale self-report version, the 28-item Mobility Inventory, the 16-item Penn State Worry Questionnaire, the 10-item Yale-Brown Obsessive Compulsive Scale self-report version, the 20-item PTSD checklist for the DSM-5, or the 14-item Whitely Index. Higher scores indicate higher symptom severity. Z-scores will be calculated from individual scores for group-level analyses.
Change from baseline in severity of depressive symptoms at post-treatment | baseline and 3 or 6 months
  Severity of depressive symptoms are measured with the 30-item Inventory for Depressive Symptomatology self-report questionnaire. Higher scores indicate higher symptom severity.
Change from baseline in severity of depressive symptoms at 3 months | baseline and 3 months
  Severity of depressive symptoms are measured with the 30-item Inventory for Depressive Symptomatology self-report questionnaire. Higher scores indicate higher symptom severity.
Change from baseline in severity of depressive symptoms at 12 months | baseline and 12 months
  Severity of depressive symptoms are measured with the 30-item Inventory for Depressive Symptomatology self-report questionnaire. Higher scores indicate higher symptom severity.
Remission rates from anxiety-related disorder at post-treatment | 3 or 6 months
  Remission of diagnoses of anxiety-related disorders is assessed using the Mini International Neuropsychiatric Interview - Simplified for DSM-5, Dutch version 1.1 (Overbeek & Schruers, 2019).
Remission rates from anxiety-related disorder at 12 months | 12 months
  Remission of diagnoses of anxiety-related disorders is assessed using the Mini International Neuropsychiatric Interview - Simplified for DSM-5, Dutch version 1.1 (Overbeek & Schruers, 2019).
New-onset anxiety-related or depressive disorder post-treatment | baseline, 3 or 6 months
  The new onset of anxiety-related or depressive disorder between baseline and post-treatment is assessed using the Mini International Neuropsychiatric Interview - Simplified for DSM-5, Dutch version 1.1 (Overbeek & Schruers, 2019)
New-onset anxiety-related or depressive disorder at 12 months | 12 months
  The new onset of anxiety-related or depressive disorder between baseline and post-treatment is assessed using the Mini International Neuropsychiatric Interview - Simplified for DSM-5, Dutch version 1.1 (Overbeek & Schruers, 2019)
Productivity costs over 12 months | 3months, 6months, 12 months
  Productivity losses are assessed using the iMTA Productivity Cost Questionnaire (iPCQ). The iPCQ is a 12-item self-report questionnaire including three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work in the past 3 months.
Medical costs over 12 months | 3months, 6months, 12 months
  Medical costs from a mental health care perspective are assessed using the iMTA Medical Cost Questionnaire (iMCQ). The iMCQ is a 23-item self-report questionnaire, which apart from some general questions include questions on medical consumption from different healthcare providers in the past 3 months.
Change from baseline in health-related quality of life over 12 months | baseline, 2 weeks, 4 weeks, 2 months, 3 months, 6 months, 12 months
  Quality of life is measured using the EQ-5D-5L. The EQ-5D-5L scores (reflecting the level of perceived problems on the dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression) are used to calculate utilities using the Dutch tariff. Quality Adjusted Life Years are calculated using linear interpolation between time points. Higher QALY scores indicate more improvement in quality of life.
Drop-out rates at post-treatment | 3 or 6 months
  Percentage of patiënts who missed more than 25% of CBT sessions.
Patient satisfaction at post-treatment | 3 or 6 months
  The 8-item Client Satisfaction Questionnaire (CSQ-8) measures overall satisfaction of the patient with health and human services. Each item on the CSQ-8 is scored from 1 (low satisfaction) to 4 (high satisfaction), possible total scores ranging 8-32.
Negative effects of psychotherapy | 3 or 6 months
  The 21-item Inventory for the Assessment of Negative Effects of Psychotherapy (INEP) is a self-report instrument for assessing negative effects of psychotherapy from the patient's perspective. The negative effects cover 7 domains: Intrapersonal Change, Intimate Relationships, Stigmatization, Emotions, Workplace, Family and Friends, and Therapeutic Malpractice. The INEP items are answered using a 4-stage response format (0 = "disagree/not applicable"; 3 = "fully agree").

CONTACTS AND LOCATIONS:
Overall Officials: Neeltje Batelaan, PhD, Study Director — Amsterdam UMC
Locations (6):
- Netherlands (6):
  - GGZ inGeest, polikliniek Angst & Dwang, locatie Amstelmere, Amstelveen
  - GGZ inGeest, polikliniek Angst & Dwang, locatie De Nieuwe Valerius, Amsterdam
  - GGZ inGeest, polikliniek Angst & Dwang, locatie Zuiderpoort, Haarlem
  - GGZ Centraal, Algemeen Specialistische Polikliniek, Hilversum
  - GGZ inGeest, polikliniek Angst & Dwang, locatie Spaarnepoort, Hoofddorp
  - Altrecht Academisch Angstcentrum, Utrecht

IPD SHARING:
Plan to Share IPD: No